CLINICAL TRIAL: NCT06669806
Title: A Prospective, Multi-Center, Single-Arm Clinical Study to Evaluate the Effectiveness and Safety of LIVERTYTM TIPS Stent Graft in the Treatment of Cirrhosis and Complications of Portal Hypertension
Brief Title: Effectiveness and Safety of TIPS Stent Graft in the Treatment of Cirrhosis and Complications of Portal Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDPI-22CHTIPS
Record Dates: First submitted 2024-10-18; First posted 2024-11-01 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Portal Hypertension Related to Cirrhosis; Ascites Hepatic; Variceal Bleeding
Keywords: Transjugular intrahepatic portosystemic shunt; TIPS stent; patency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TIPS Stent Graft device (Experimental): after creating and dilating the hepatic parenchymal tract, the device is planted to cover the intrahepatic shunt and hepatic vein. A second stent graft may be placed in overlapped fashion.
  Interventions: Device: TIPS Stent Graft

INTERVENTIONS:
Device: TIPS Stent Graft — a covered TIPS stent graft

SUMMARY:
This Study is a prospective, multi-center, single-arm objective perform an criteria (OPC) study. A 12 months follow-up study on the patients who intend to receive the treatment of cirrhosis and complications of portal hypertension with the TIPS Stent Graft will be conducted. The primary evaluation endpoint of this Study is the stent patency at 6 months after treatment completion .

ELIGIBILITY:
Inclusion Criteria:

1. The subject who is 18 years old or above but 75 years old or below;
2. The subject who is diagnosed with portal hypertension caused by liver cirrhosis with the history of gastrointestinal variceal bleeding or bleeding, hepatic hydrothorax, and refractory or recurrent ascites;
3. The subject must have adequate functional hepatic reserve with a Model for End-Stage Liver Disease (MELD) Score of ≤13 or Child-Pugh Score of ≤18;
4. The subject with platelet count≥ 20×10^9 /L;
5. Subjects or their guardians who can understand the content of the clinical trial, voluntarily participate in the clinical trial and sign the ICF and can complete the follow-up period according to the requirements of the clinical trial.

Exclusion Criteria:

1. The subject who is pregnant or lactating or plan to get pregnant during the clinical trial;
2. According to the judgment of investigator, the subject with main portal vein thrombosis which thrombus occupying >50% of the portal vein lumen and affecting postoperative hemodynamics;
3. The subject who has received surgical or interventional treatment (such as TIPS, surgical shunt and retrograde transvenous obliteration (-RTO) for treatment of complications from portal hypertension. Note: The subject who have received -RTO for variceal bleeding at least 8 weeks before signing the informed consent form can be included in the clinical trial;
4. The subject who needs to receive or have received splenectomy;
5. The subject who has received or plan to receive liver transplantation;
6. The subject who cannot have a shunt channel established in the liver parenchyma between the hepatic vein and the portal vein as determined by the investigators;
7. The subject with extrahepatic or hepatic malignancies;
8. The subject with Budd-Chiari syndrome and hepatic sinusoidal obstruction syndrome;
9. The subject with congenital cystic dilatation of bile duct (Caroli disease) and obstructive dilation of biliary tract;
10. The subject with polycystic liver disease;
11. The subject with cavernous transformation of the portal vein;
12. The subject with severe or refractory hepatic encephalopathy (Grade 2 or above according to the West Haven Criteria);
13. The subject with a TBIL level higher than 51.3 μmol/L (excluding the Patients with cholestatic cirrhosis);
14. The subject with coagulation disorders (INR: >2.5);
15. The subject with a systolic pressure lower than 80 mmHg;
16. The subject with severe tricuspid regurgitation or congestive heart failure;
17. The subject with myocardial infarction within the past 3 months;
18. The subject with moderate to severe pulmonary arterial hypertension, or severe hepatopulmonary syndrome;
19. The subject with uncontrolled systemic infection or inflammation;
20. The subject with severe renal insufficiency (Scr level:>199.5 μmol/L) or needing to receive dialysis;
21. The subject known to be allergic to the contrast media or to the constituent materials of the TIPS covered segment;
22. The subject with the history of epilepsy or mental illness or with cognitive impairment;
23. The subject with the expected survival time of less than 1 year;
24. The subject who is otherwise determined as ineligible for participation in this Study by investigators;
25. The subject who is participating in any other unfinished drug or medical device clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Stent patency rate after treatment completion* | 6 months

SECONDARY OUTCOMES:
Technical success rate | immediately after the intervention
Hemodynamic success rate | immediately after the intervention
Incidence of subjects free from receiving TIPS shunt reoperation after treatment completion* | 1 month, 3 months, 6 months and 12 months
Stent patency rate after treatment completion* | 1 month, 3 months and 12 months
Incidence of subjects free from severe hepatic encephalopathy after treatment completion* | 1 month, 3 months, 6 months and 12 months
Incidence of subjects free from rebleeding after treatment completion* | 1 month, 3 months, 6 months and 12 months
The proportion of clinical improvement on ascites after treatment completion* | 3 months, 6 months, and 12 months
The proportion of clinical improvement on hepatic hydrothorax after treatment completion* | 3 months, 6 months, and 12 months
Liver transplant-free survival rate post-index procedure | 6 months and 12 months
Overall survival rate post-index procedure | 1 month, 3 months, 6 months and 12 months
Incidence of medical device-related and/or operation-related severe complications | 1 month
TEP related adverse events (AE) after treatment completion* | 6 months and 12 months
Adverse events (AE) after index procedure | 6 months and 12 months
Serious adverse events (SAE) after index procedure | 6 months and 12 months
Device deficiencies | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial People's Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No